CLINICAL TRIAL: NCT06842498
Title: A Phase 2 Dose Optimization Trial Evaluating a CD46-Targeted Antibody-Drug Conjugate (FG-3246) in Patients With Metastatic Castration-Resistant Prostate Cancer
Brief Title: A Study of FG-3246 in Participants With Metastatic Castration-Resistant Prostate Cancer (mCRPC)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kyntra Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FGCL-3246-112
Record Dates: First submitted 2025-02-19; First posted 2025-02-24 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Castration-Resistant Prostate Cancer
Keywords: FG-3246; FOR46; mCRPC; CRPC; CD46; Prostate cancer; Antibody-drug conjugate; Metastatic prostate cancer; FibroGen; ADC
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- FG-3246 1.8 mg/kg (Experimental): Participants will receive FG-3246 1.8 milligrams (mg)/kilogram (kg) administered via intravenous (IV) infusion on Day 1 of each 21-day treatment cycle (every 3 weeks [Q3W]) until radiographic progression, unacceptable safety and tolerability, participant or investigator decision to stop treatment, other withdrawal criteria are met, or FibroGen decision to close the study.
  Interventions: Drug: FG-3246
- FG-3246 2.4 mg/kg (Experimental): Participants will receive FG-3246 2.4 mg/kg administered via IV infusion on Day 1 of each 21-day treatment cycle (Q3W) until radiographic progression, unacceptable safety and tolerability, participant or investigator decision to stop treatment, other withdrawal criteria are met, or FibroGen decision to close the study.
  Interventions: Drug: FG-3246
- FG-3246 2.7 mg/kg (Experimental): Participants will receive FG-3246 2.7 mg/kg administered via IV infusion on Day 1 of each 21-day treatment cycle (Q3W) until radiographic progression, unacceptable safety and tolerability, participant or investigator decision to stop treatment, other withdrawal criteria are met, or FibroGen decision to close the study.
  Interventions: Drug: FG-3246

INTERVENTIONS:
Drug: FG-3246 — FG-3246 will be administered per schedule specified in the arm description.
  Other Names: FOR46

SUMMARY:
The purpose of this study is to evaluate the safety, efficacy, tolerability, and pharmacokinetics (PK) of FG-3246, a cluster of differentiation 46 (CD46) targeting antibody-drug conjugate (ADC), in the treatment of participants with mCRPC who have progressed following treatment with one prior second-generation androgen receptor signaling inhibitor (ARSI) in any setting and no prior taxane therapy in the mCRPC setting.

ELIGIBILITY:
Key Inclusion Criteria:

* Participant must have histological, and/or cytological confirmation of prostate adenocarcinoma.
* Participant with safely accessible tumor lesion must agree to biopsy of a primary or metastatic lesion during screening. Alternatively, participant may provide an archival biopsy of a primary or metastatic lesion that was taken after castration resistance developed and within 1 year prior to randomization.
* Participant must have serum testosterone levels <50 nanograms (ng)/deciliter (dL) during screening.
* Participant is required to have progressed on one prior treatment with a second generation ARSI (abiraterone acetate, enzalutamide, apalutamide, or darolutamide) initiated in either the castration-sensitive or castration-resistant setting.
* Participant must have progressive mCRPC following last treatment at screening.
* Participant must have ≥1 metastatic lesion that is present on baseline Computed Tomography (CT), Magnetic Resonance Imaging (MRI), or bone scan obtained ≤28 days prior to randomization.
* Participant must have adequate organ function during screening and reconfirmed on Study Day -1 or Day 1.

Key Exclusion Criteria:

* Participant has received previous treatment with a therapeutic targeting CD46.
* Participant has small cell neuroendocrine carcinoma (pure or mixed) or any other non-adenocarcinoma component on prior or current histologic evaluation of primary or metastatic lesion.
* Participant has received more than one prior second-generation ARSI in any setting.
* Participant has received any systemic anticancer therapy (for example, hormonal therapy, chemotherapy, immunotherapy, radioligand therapy, or biological therapy [including monoclonal antibodies], including investigational therapy) within 28 days prior to randomization.
* Participant has received any prior radiation therapy within 28 days prior to randomization.
* Participant has a known actionable mutation or gene alteration, for example, BRCA1 mutation, for which approved therapies are available, for example, PARP inhibitors, unless these therapies are not appropriate for the participant as determined by the investigator or the participant refuses such therapy.
* Participant has National Cancer institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) ≥Grade 2 peripheral neuropathy at the time of screening from any etiology.
* Participant has received any prior chemotherapy; however, one prior taxane-based chemotherapy in the castration-sensitive setting is allowed if completed >12 months before randomization.
* Participant has known hypersensitivity to the components of FG-3246 or its analogs or a history of allergic or anaphylactic reaction to human, humanized, or chimeric monoclonal antibodies.
* Participant has diagnosis with any other malignancy in the past 5 years, except for adequately treated basal cell or squamous cell carcinoma of the skin.
* Participant requires treatment with a strong cytochrome P450 3A4 (CYP3A4) inhibitor or inducer drug that cannot be safely discontinued.

NOTE: Other protocol-defined inclusion/exclusion may apply.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Radiographic Progression-free Survival (rPFS) By Investigator Assessment Per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and Prostate Cancer Clinical Trials Working Group 3 (PCWG3) Criteria | Until radiographic progression is noted (up to approximately 30 months)
Number of Participants With Treatment-emergent Adverse Events (TEAEs) | From first dose until 28 days after last dose (up to approximately 30 months)
Maximum Plasma Concentration (Cmax) of FG-3246, Total Anticluster of Differentiation 46 Antibody (CD46), and Free Monomethyl Auristatin E (MMAE) | Within each 21 day treatment cycle from Cycle 1 through 28 days post last dose (up to approximately 30 months)

SECONDARY OUTCOMES:
rPFS Rate at 6 Months (rPFS6) Per RECIST v1.1 and PCWG3 Criteria | Month 6
rPFS Rate at 12 Months (rPFS12) Per RECIST v1.1 and PCWG3 Criteria | Month 12
Confirmed Objective Response Rate (ORR) Per RECIST v1.1 and PCWG3 Criteria | From first dose up to approximately 30 months
Duration of Response (DoR) Per RECIST v1.1 and PCWG3 Criteria | From first dose up to approximately 30 months
Confirmed PSA50 Response Rate: Percentage of Participants Achieving a Decline in Prostate-specific Antigen (PSA) ≥50% From Baseline | Up to approximately 30 months
Confirmed PSA90 Response Rate: Percentage of Participants Achieving a Decline in PSA ≥90% From Baseline | Up to approximately 30 months
Composite Response Rate (CRR) Per RECIST 1.1 and PCWG3 Criteria | Up to approximately 30 months
PSA Progression-free Survival (PFS) | Up to approximately 30 months
Disease Control Rate (DCR) per RECIST 1.1 and PCWG3 Criteria | Up to approximately 30 months
Clinical Benefit Rate (CBR) per RECIST 1.1 and PCWG3 Criteria | Up to approximately 30 months
Time to First Symptomatic Skeletal-related Event (SSRE) | Up to approximately 30 months
Overall Survival (OS) | Until death or up to approximately 30 months
Percentage of Participants Who Develop Antidrug Antibodies (ADA) and Neutralizing Antibody (NAb) Against FG-3246 | Within each 21 day treatment cycle from Cycle 1 through 28 days post last dose (up to approximately 30 months)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - The University of Arizona Cancer Center - North Campus, Tucson, Arizona
  - UCLA Clark Urology Center, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - Bioresearch Partner, Aventura, Florida
  - Bioresearch Partner, Hialeah, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - UNC Hospitals, The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center - Duke Cancer Center, Durham, North Carolina
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Oncology Consultants, Houston, Texas
  - University of Virginia Comprehensive Cancer Center, Charlottesville, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington